CLINICAL TRIAL: NCT03604965
Title: A Multicenter, Randomized Controlled Phase III Clinical Trial of GP Induction Chemotherapy With TPF Adjuvant Chemotherapy Combined With DDP Concurrent Chemoradiotherapy in the Treatment of Locally Advanced Nasopharyngeal Carcinoma
Brief Title: GP Induction Chemotherapy us TPF Adjuvant Chemotherapy Combined With DDP Concurrent Chemoradiotherapy in the Treatment of Locally Advanced NPC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guiyang Medical University (Other)
Responsible Party: Principal Investigator, Feng Jing, Head and neck cancer director, chief researcher, clinical professor, Guiyang Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201805043
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP+CCRT (Experimental): GP neoadjuvant chemotherapy followed by cisplatin chemotherapy concurrent combined with intensity-modulated radiation therapy
  Interventions: Drug: GP+CCRT
- TPF+CCRT (Active Comparator): TPF neoadjuvant chemotherapy followed by cisplatin chemotherapy concurrent combined with intensity-modulated radiation therapy
  Interventions: Drug: TPF+CCRT

INTERVENTIONS:
Drug: GP+CCRT — Patients receive Neoadjuvant gemcitabine (1000mg/m2 on day1 and day8 ) and cisplatin (80mg/m2 on day1)every 21days for three cycles followed by concurrent cisplatin (100mg/m2 on day1 or day2)every 21 days for three cycles during radiotherapy
  Other Names: Experimental group
  Arms: GP+CCRT
Drug: TPF+CCRT — Patients receive Neoadjuvant Docetaxel (75mg/m2 on day1 03:30-04:30) and cisplatin (75mg/m2 on day 1-5 10:00-22:00) and 5-FU(750mg/m2 on day 1-5 22:00-10:00) every 21days for three cycles followed by concurrent cisplatin (100mg/m2 on day1 or day2)every 21 days for three cycles during radiotherapy
  Other Names: Control group
  Arms: TPF+CCRT

SUMMARY:
Through randomized controlled phase III multicenter clinical trials, GP induction chemotherapy vs TPF regimen adjuvant chemotherapy combined with DDP concurrent chemoradiotherapy for the treatment of locally advanced nasopharyngeal carcinoma: the efficacy, toxicity and quality of life, and further improvement Survival rate and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. In the newly diagnosed patient, no radiotherapy or chemotherapy was performed before the start of the clinical trial.
2. Pathologically confirmed as non-keratinizing nasopharyngeal carcinoma (differentiated or undifferentiated, ie WHO type II or III).
3. III, IVa patients (AJCC version 8 staging).
4. Male or non-pregnant women.
5. Age ≥ 18 and < 70 years old.
6. Functional status: Karnofsky scale (KPS) > 70.
7. White blood cells (WBC) ≥ 4 × 109.

   /L, hemoglobin (HGB) ≥ 90 g / L, platelets (PLT) ≥ 100 × 109 / L (or within the normal range of the laboratory)
8. Liver function: alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 1.5 times the upper limit of normal (ULN); Total bilirubin ≤ 1.5 × ULN.
9. Renal function: creatinine clearance ≥ 60ml / min or serum creatinine ≤ 1.5 × ULN.
10. The patient has signed an informed consent form.

Exclusion Criteria:

1. The pathological type is WHO's keratinized squamous cell carcinoma or basal squamous cell carcinoma.
2. Age ≥ 70 years old or < 18 years old.
3. Treatment is palliative.
4. Previous history of malignant tumors, well-treated basal cell carcinoma or squamous cell carcinoma and cervical carcinoma in situ outer.
5. Women during pregnancy or lactation (pregnant women should be considered for women of childbearing age; Effective contraception).
6. Previously received radiation therapy (if non-melanoma skin cancer and previous lesions are outside the target area of radiotherapy, then except).
7. Primary and cervical metastatic lesions received chemotherapy or surgery (except for diagnostic treatment).
8. With other serious diseases, it may bring greater risk or affect the compliance of the test. For example: no need for treatment Stable heart disease, kidney disease, chronic hepatitis, control of unsatisfactory diabetes (fasting blood glucose > 1.5 × ULN),And mental illness.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2018-07-21 (Actual); Primary Completion 2020-07-21 (Estimated); Study Completion 2020-07-21 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | 3 years
  Progress-free survival(year) is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  The OS(year) was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional failure-free survival(LRFS) | 3 years
  The LRFS(year) is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant metastasis-free survival(DMFS) | 3 years
  The DMFS(year) is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Overall response rate | 3 years
  Tumour response(CR/PR/SD/PD) was classified according to RECIST v1.1
Incidence of acute and late toxicity | 3 years
  Incidence of acute toxicity（Grade1/2/3/4） is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme

CONTACTS AND LOCATIONS:
Overall Officials: Yuanyuan Li, Master, Principal Investigator — Guizhou Provincial Cancer Hospital
Locations (1):
- Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No